CLINICAL TRIAL: NCT04893252
Title: Vactosertib in Combination With Durvalumab (MEDI4736) in Patients With Gastric Cancer
Brief Title: Vactosertib and Durvalumab in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hark Kyun Kim (Other Government)
Responsible Party: Sponsor-Investigator, Hark Kyun Kim, Principle Investigator, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33737
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — durvalumab; vactosertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vactosertib in combination with durvalumab (Experimental): single arm study
  Interventions: Drug: durvalumab and vactosertib

INTERVENTIONS:
Drug: durvalumab and vactosertib — durvalumab IV Q4W in combination with vactosertib PO bid (5 days a week)

SUMMARY:
This trial will test the efficacy and safety of durvalumab in combination with vactosertib in patients with metastatic gastric cancers who failed ≥ 2 lines of chemotherapy

DETAILED DESCRIPTION:
Efficacy and safety of durvalumab (anti-PD-L1) via IV infusion Q4W, in combination with vactosertib (TGF-beta inhibitor) PO bid for 5 days a week for up to a maximum of 12 months, will be tested in patients with metastatic hypermutated gastric cancers as ≥ 3rd-line setting until confirmed disease progression, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically- or cytologically-confirmed diagnosis of metastatic gastric adenocarcinoma in the stomach and gastroesophageal junction that are refractory to at least two lines of treatment.
* Have a performance status of 0-1 on the ECOG Performance Scale.
* Have measurable disease at least one investigator-assessed measurable disease per RECIST v1.1
* Have adequate organ functions

Exclusion Criteria:

* Prior ALK5 inhibitor treatment
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study drugs
* Patients weighing <30kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Every 8 weeks from the date of the first dose until the date of progression, assessed up to 1 year
  Objective response rate in 55 participants according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No